CLINICAL TRIAL: NCT06859411
Title: Prognosis of Posterior Lamellar Keratoplasty: an Observational Cohort Study
Brief Title: Prognosis of Posterior Lamellar Keratoplasty, an Observational Cohort Study
Acronym: CORNEACOHORT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-11Obs-CHRMT
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Fuchs' Endothelial Corneal Dystrophy; Pseudophakic Bullous Keratopathy
Keywords: posterior lamellar keratoplasty; cornea; DMEK; DSAEK
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DMEK: Patients who received Descemet Membrane Endothelial Keratoplasty
  Interventions: Procedure: visual acuity comparaison
- DSAEK: Patients who received Descemet Stripping Automated Endothelial Keratoplasty with preoperative graft thicker than 160 µm
  Interventions: Procedure: visual acuity comparaison
- UT-DSAEK: DSAEK: patients who received Descemet Stripping Automated Endothelial Keratoplasty with preoperative graft thinner than 160 µm
  Interventions: Procedure: visual acuity comparaison

INTERVENTIONS:
Procedure: visual acuity comparaison — Data collection

SUMMARY:
Over the past decade, the management of Fuchs' endothelial corneal dystrophy (FECD) and pseudophakic bullous keratopathy (PBK) has been revolutionized by the development of posterior lamellar keratoplasty techniques: DSAEK and DMEK.

DSAEK (Descemet Stripping Automated Endothelial Keratoplasty) involves replacing the patient's endothelium and pathological descemetum with a descemetic endothelial graft combined with a thin stromal lamella. The endothelial density of the grafts is generally greater than 2,400 cells/mm². Depending on the grafting center and tissue bank, grafts may be either pre-cut in the tissue bank or cut on the operating table by the surgeon himself.

The donor graft is placed on an artificial anterior chamber, and automated microkeratome cutting produces grafts with an average thickness of 100 to 200µm, sometimes less than 100um (known as UT-DSAEK or ultra-thin DSAEK).

DMEK (Descemet Membrane Endothelial Keratoplasty) is a strictly endothelium and Descemet's membrane graft, as close as possible to the original anatomy of the cornea. The graft is dissected manually either in a tissue bank (pre-cut grafts) or on the operating table by the surgeon. The thickness of the graft is between 15 and 18 microns.

The primary objective of this observational cohort is to compare the evolution of visual acuity after DMEK, DSAEK or UT-DSAEK transplantation.

Secondary objectives are to compare the evolution of endothelial cell density, corneal thickness and early and late post-operative complications, and to identify factors predictive of these different endpoints.

ELIGIBILITY:
Inclusion Criteria:

* patients who received a posterior lamellar keratoplasty in Metz-Thionville Regional Hospital between 2012 and 2030

Exclusion Criteria:

* patients refusing to take part in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who received a posterior lamellar keratoplasty
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2040-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
BSCVA | at 1 year after surgery, but also at day 8, day 15, 1 month, 3 months, 6 months and every year up to 10 years after surgery
  best spectacle-corrected visual acuity (logMAR)

SECONDARY OUTCOMES:
ECD | at 1 month, 3 months, 6 months and every year up to 10 years after surgery
  endothelial cell count (cells/mm²)
CCT | at 1 month, 3 months, 6 months and every year up to 10 years after surgery
  central cornea thickness (µm)
post-operative complication | up to 10 years after surgery
  graft reject (yes/no), graft detachment (yes/no), graft failure (yes/no), eye infection (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc PERONE, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No
No
  According to the French law and the French Data Protection Authority (CNIL), we won't be able to publicly share individual participant data, but we plan to share their conclusions through peer-reviewed publications and conferences.